CLINICAL TRIAL: NCT05373927
Title: Cross-sectional Study of Calf Muscle Perfusion in Patients With Intermittent Claudication by Non-invasive Multispectral Optoacustic Tomography
Brief Title: Calf Muscle Perfusion in Patients With Intermittent Claudication by Non-invasive MSOT
Acronym: MSOT_IC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ulrich Rother (Other)
Collaborators: PD Dr. med. Ferdinand Knieling, Department of pediatrics, University of Erlangen-Nürnberg (Unknown)
Responsible Party: Sponsor-Investigator, Ulrich Rother, PD Dr. med., University Hospital Erlangen
Organization: University Hospital Erlangen (Other)
Other Study IDs: MSOT_IC
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Vascular Diseases; Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Artery Disease; PAD; Intermittent Claudication; Claudicatio intermittens; Critical Limb Ischaemia; CLI; Critical Limb Threatening Ischemia; CTLI; Color-Coded Duplex Sonography; CCDS; Ankle Brachial Index; ABI; Multispectral Optoacoustic Tomography; MSOT; Heel Raises; 6-minute walk test; 6MWT; Muscle Perfusion; Calf Muscle Perfusion
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group 1: Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus triceps surae of the affected leg in PAD patients in Fontaine stage II (intermittent claudication) or one leg in healthy volunteers (total 1 site)
  Physical assessment: Pulse status / Color-Coded Duplex Sonography / Ankle-Brachial Index / 6-minute walk test (6MWT) / Continued heel raises for at least 30s
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Study group 2: Multispectral Optoacoustic Tomography (MSOT) and B-Mode Ultrasound of the Musculus triceps surae of the affected leg in PAD patients in Fontaine stage II (intermittent claudication) or one leg in healthy volunteers (total 1 site)
  Physical assessment: Pulse status / Color-Coded Duplex Sonography / Ankle-Brachial Index / 6-minute walk test (6MWT) / Continued heel raises for at least 30s
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous imaging of subcellular muscle components via infrared and near-infrared laser pulses

SUMMARY:
The objective of the proposed study is to define independent parameters for the diagnostic assessment of the perfusion situation of the calf muscle based on multispectral optoacoustic tomography (MSOT) in a cross-sectional collective of patients with PAD in Fontaine stage II (intermittent claudication) and a healthy control collective (study group 1). The results will be validated using an independent validation group (study group 2).

DETAILED DESCRIPTION:
PAD is one of the most common diseases of the elderly. As life expectancy increases, there is a growing need for new treatment concepts and new diagnostic procedures.

Up to now, only the measurement of macrocirculation in the form of CCDS, ABI and measurement of the actual walking distance are available as independent validation measures of revascularization methods (endovascular/open). The S3 guideline for diagnosis, therapy and medical aftercare of PAD published in 2015 by DGA (Deutsche Gesellschaft für Angiologie, German Society for Angiology) recommends such aftercare examinations, especially for patients that underwent vascular surgery. However, for the mentioned validation measures there are some patient groups for which these methods provide only insufficient or unusable results (e.g. diabetes mellitus, terminal renal failure). In these cases, independent verification of the success of the chosen therapy would have to be performed using angiography (digital subtraction angiography, CT angiography or MR angiography). However, this is not routinely performed in the respective patient populations due to the associated risks (including radiation exposure, contrast agent administration, invasiveness).

MSOT provides a new non-invasive diagnostic method that may be able to fill this diagnostic gap. A first study (MSOT_PAD, NCT04641091) confirmed the hypothesis that data collected via MSOT examination of the calf muscle can be used for PAD diagnostics. The derived concentration of oxygenated hemoglobin (HbO2) proved to be the most suitable measurement parameter. A connection could be established between the measured HbO2 concentration and the clinical stage of PAD. Differentiation improved after a standardized exercise of a walking distance of 150 meters, with patients in the stage of intermittent claudication (IC, Fontaine stage II) being more difficult to differentiate in comparison to patients in Fontaine stages III and IV.

The aim of this cross-sectional study is to increase the sensitivity and specificity of the procedure for IC patients by using a more suitable exercise between first and second MSOT measurement, namely repeated heel raises until the occurrence of claudication pain. A subgroup of the IC patients having been included in the study will be asked to undergo the study protocol a second time after interventional/ surgical revascularization. This is to investigate whether and how the improved blood flow situation translates to the measured MSOT parameters.

As additional target variables, the relative, absolute and total walking distance in a 6-minute walk test as well as the PAD-specific quality of life will be recorded with the VASCUQOL-6 questionnaire. A healthy control collective is included as a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with manifest PAD in stage II according to Fontaine or categories 1-3 according to Rutherford or healthy volunteers
* Adults (>18 years) who are able to give their consent

Exclusion Criteria:

* Patients with PAD stage I, III and IV according to Fontaine or categories 0, 4, 5 and 6 according to Rutherford or healthy volunteers with diabetes mellitus, chronic renal failure, claudication symptoms, abnormal ABI or non-palpable foot pulses
* Underage persons
* Lack of written consent
* Safety concerns of the study physician (person with physical, mental or psychiatric conditions which, by the judgement of the study physician, would compromise the person's safety or the quality of the data, thereby rendering the person an ineligible candidate for the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with
  * PAD IIa
  * PAD IIb presenting for consultation during consultation hours of the department of vascular surgery.
  Healthy volunteers being recruited by notices posted in the clinic with following conditions:
  * no PAD previously known
  * no diabetes mellitus previously known
  * no chronic renal insufficiency previously known
  * no symptoms of intermittent claudication
  * ABI with values between 0.9 and 1.4 (screening examination before inclusion in the study)
  * palpable foot pulses
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Optimal diagnostic MSOT thresholds | single time point (1 day)
  Optimal diagnostic threshold for hemoglobin-associated MSOT parameters in calf muscle tissue in patients with intermittent claudication before and after exercise

SECONDARY OUTCOMES:
Difference between the corresponding MSOT values before and after exercise | single time point (1 day)
  Difference of the values before and after exercise for hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with IC
Reperfusion profiles for hemoglobin-associated parameters | single time point (1 day)
  Curves of hemoglobin-associated MSOT parameters in the first ten minutes after exercise
Correlation of acquired MSOT parameters with the CCDS flow profile and PSV | single time point (1 day)
  Hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) in patients with IC correlated with the flow profile and PSV of A. femoralis communis and A. poplitea determined by CCDS
Correlation of acquired MSOT parameters with the ABI | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the ABI
Correlation of acquired MSOT parameters with relative and absolute walking distance | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with relative (until the first occurrence of pain) and absolute walking distance (until the first stopping due to pain) in the 6-minute walk test (6MWT)
Correlation of acquired MSOT parameters with maximum walking distance within 6 minutes | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the maximum walking distance during the 6 minutes of the 6-minute walk test
Correlation of acquired MSOT parameters with the subjectively perceived maximum walking distance in everyday life | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the subjectively perceived maximum walking distance in everyday life
Correlation of acquired MSOT parameters with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire) | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT correlated with the perceived PAD-specific quality of life (VASCUQOL-6 questionnaire)
Correlation of the acquired MSOT parameters with the TASC-classification (angiography) | single time point (1 day)
  Hemoglobin-associated parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with IC correlated with the TASC-classification (angiography) [If angiographic imaging is already available due to routine diagnostics independently from this study.]
Subgroup analysis: Difference between the corresponding MSOT values before and after revascularization intervention | two time points (2 days)
  Subgroup analysis: Difference of the MSOT values before and after revascularization intervention for hemoglobin-associated parameters derived by transcutaneous MSOT in patients with IC
Subgroup analysis: Reperfusion profiles for hemoglobin-associated parameters after revascularization intervention | single time point (1 day)
  Subgroup analysis: Reperfusion profiles of hemoglobin-associated MSOT parameters (i.e. the curves of hemoglobin-associated MSOT parameters in the first ten minutes after exercise) after revascularization intervention
Subgroup analysis: Correlation of acquired MSOT parameters after intervention with the CCDS flow profiles and PSVs after intervention | single time point (1 day)
  Subgroup analysis: hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT in patients with IC after revascularization intervention correlated with the flow profiles and PSVs of A. femoralis communis and A. poplitea determined by CCDS after revascularization intervention
Subgroup analysis: Correlation of acquired MSOT parameters after intervention with the ABI after intervention | single time point (1 day)
  Subgroup analysis: hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT after revascularization intervention correlated with the ABI measurements after revascularization intervention
Subgroup analysis: Correlation of acquired MSOT parameters after intervention with relative (until the first occurrence of pain) and absolute walking distance (until the first stopping due to pain) determined during the 6MWT after intervention | single time point (1 day)
  Subgroup analysis: hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT after revascularization intervention correlated with relative (until the first occurrence of pain) and absolute walking distance (until the first stopping due to pain) in the 6MWT after revascularization intervention
Subgroup analysis: Correlation of acquired MSOT parameters after intervention with maximum walking distance in the 6MWT after intervention | single time point (1 day)
  Subgroup analysis: hemoglobin-associated MSOT parameters (units: arbitrary units (a.u.)) derived by transcutaneous MSOT after revascularization intervention correlated with the maximum walking distance in the 6MWT after revascularization intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Erlangen-Nuremberg (FAU), Department of Vascular Surgery, Erlangen, Bavaria, Germany

REFERENCES:
- [Background] Lawall H, Diehm C, Hoffmann U, Reinecke H. [Update PAVK: Epidemiology, comorbidity and prognosis of peripheral arterial obstructive disease]. Dtsch Med Wochenschr. 2015 Dec;140(24):1798-802. doi: 10.1055/s-0041-107064. Epub 2015 Dec 1. German. PMID 26625226
- [Background] Lawall H, Huppert P, Espinola-Klein C, Zemmrich CS, Ruemenapf G. German guideline on the diagnosis and treatment of peripheral artery disease - a comprehensive update 2016. Vasa. 2017 Mar;46(2):79-86. doi: 10.1024/0301-1526/a000603. Epub 2017 Jan 27. PMID 28128018
- [Background] Alpert JS, Larsen OA, Lassen NA. Exercise and intermittent claudication. Blood flow in the calf muscle during walking studied by the xenon-133 clearance method. Circulation. 1969 Mar;39(3):353-9. doi: 10.1161/01.cir.39.3.353. No abstract available. PMID 4885945
- [Background] Karlas A, Masthoff M, Kallmayer M, Helfen A, Bariotakis M, Fasoula NA, Schafers M, Seidensticker M, Eckstein HH, Ntziachristos V, Wildgruber M. Multispectral optoacoustic tomography of peripheral arterial disease based on muscle hemoglobin gradients-a pilot clinical study. Ann Transl Med. 2021 Jan;9(1):36. doi: 10.21037/atm-20-3321. PMID 33553329
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901

DOCUMENTS (2):
  • Study Protocol (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT05373927/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT05373927/SAP_001.pdf